CLINICAL TRIAL: NCT00963950
Title: Transvaginal Cholecystectomy
Brief Title: Transvaginal Cholecystectomy Versus Laparoscopic Cholecystectomy in Patients With Biliary Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0902004771
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Biliary Colic
Keywords: cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): transvaginal cholecystectomy
  Interventions: Procedure: transvaginal cholecystectomy
- laparoscopic cholecystectomy (Active Comparator): Laparoscopic cholecystectomy (4 port)
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: transvaginal cholecystectomy — Transvaginal approach to gallbladder removal.
  Arms: Intervention group
Procedure: laparoscopic cholecystectomy — laparoscopic cholecystectomy
  Arms: laparoscopic cholecystectomy

SUMMARY:
A safe and effective transvaginal approach accessing the abdominal cavity through the vagina rather than the abdominal wall is today considered a routine approach for many gynecologic surgeries.

First described by Dr. Ott in Germany in 1901, it is used routinely for transvaginal surgery, for example, transvaginal hysterectomies. This transvaginal technique has been shown to compare favorably to a laparoscopic abdominal approach because of less postoperative pain, the total elimination of abdominal wall hernias and wound infections, earlier recovery and better cosmesis.

Although routinely used in gynecological surgery, the advantages of the vaginal approach have not been utilized for general surgery applications such as cholecystectomies. Open or laparoscopic cholecystectomy accessing the abdominal cavity through abdominal wall incisions is currently still considered the standard of care in general surgery for patients with symptomatic gallbladder disease.

The investigators intend to access the abdominal cavity through the posterior vaginal fornix instead of the transabdominal approach that is now performed routinely. So far, this method of accessing the abdominal cavity through the transvaginal approach for the purpose of performing intraabdominal general surgery.

The investigators' transvaginal approach has the strong potential to further decrease invasiveness and take minimally invasive surgery to the next level in order to benefit the patient even more by minimizing postoperative pain, eliminating the risk of abdominal hernias and wound infections, improving cosmetic appearance and enabling the patient to return to routine activity and work earlier. First preliminary studies show these advantages but further research needs to be done to confirm these early positive results.

ELIGIBILITY:
Inclusion Criteria:

* Female.
* Age between 18 and 65 years old.
* Biliary dyskinesia with documented Gallbladder EF < 30% or diagnosis of biliary colic with documented gallstones or polyps by imaging.
* Body Mass Index (BMI) < 45 kg/m2.

Exclusion Criteria:

* Any female patient, who is pregnant, suspected pregnant, or lactating.
* Any patient with acute or acalculous cholecystitis.
* Any patient with an American Society of Anesthesiologists Score > 3.
* Any patient who is undergoing Peritoneal Dialysis (PD).
* Patients who are taking immunosuppressive medications or are immunocompromised.
* Patients on blood thinners or aspirin or abnormal blood coagulation tests.
* Patients who have a history of prior open abdominal surgery or prior transvaginal surgery.
* Patients with a history of ectopic pregnancy, pelvic inflammatory disease (PID) or severe endometriosis.
* Non English speaking patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
feasibility of transvaginal cholecystectomy | 2 year

SECONDARY OUTCOMES:
pain | 2 years
quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Roberts, MD, Principal Investigator — Yale University

REFERENCES:
- [Derived] Solomon D, Shariff AH, Silasi DA, Duffy AJ, Bell RL, Roberts KE. Transvaginal cholecystectomy versus single-incision laparoscopic cholecystectomy versus four-port laparoscopic cholecystectomy: a prospective cohort study. Surg Endosc. 2012 Oct;26(10):2823-7. doi: 10.1007/s00464-012-2253-0. Epub 2012 May 2. PMID 22549370